CLINICAL TRIAL: NCT07120555
Title: Outcomes of Atherectomy and Balloon Angioplasty Compared to Conventional Angioplasty in Infra-popliteal Chronic Limb-Threatening Ischemia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Moustafa Farouk, assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DFGCUOHBTR
Record Dates: First submitted 2025-07-16; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Chronic Limb Threatening Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia | interventions — Atherectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- atherectomy + balloon angioplasty (Experimental)
  Interventions: Device: atherectomy
- conventional balloon angioplasty (Experimental)
  Interventions: Device: Percutaneous transluminal angioplasty of infra-popliteal arteries lesions with primary long

INTERVENTIONS:
Device: atherectomy — Conventional balloon angioplasty remains a first-line endovascular treatment but is limited by high restenosis and vessel recoil rates. Atherectomy, a plaque debulking technique, aims to improve luminal gain and vessel compliance prior to angioplasty, potentially enhancing outcomes in heavily calcified lesions. The combination of atherectomy and balloon angioplasty has shown promise in reducing dissection rates and improving technical success, yet its superiority over conventional angioplasty alone remains controversial.
  Arms: atherectomy + balloon angioplasty
Device: Percutaneous transluminal angioplasty of infra-popliteal arteries lesions with primary long — Percutaneous transluminal angioplasty of infra-popliteal arteries lesions with primary long
  Arms: conventional balloon angioplasty

SUMMARY:
Chronic limb-threatening ischemia (CLTI) represents the most advanced stage of peripheral artery disease (PAD), characterized by rest pain, non-healing ulcers, or gangrene, and is associated with high morbidity and risk of amputation if left untreated. Infra-popliteal arteries are frequently involved in CLTI, especially in diabetic and elderly patients, posing significant challenges due to diffuse, calcified, and long-segment occlusive lesions.

Conventional balloon angioplasty remains a first-line endovascular treatment but is limited by high restenosis and vessel recoil rates. Atherectomy, a plaque debulking technique, aims to improve luminal gain and vessel compliance prior to angioplasty, potentially enhancing outcomes in heavily calcified lesions. The combination of atherectomy and balloon angioplasty has shown promise in reducing dissection rates and improving technical success, yet its superiority over conventional angioplasty alone remains controversial.

Given the growing use of endovascular therapies, a comparative analysis of outcomes between combined atherectomy-balloon angioplasty and conventional angioplasty in infra-popliteal interventions is essential to guide evidence-based management in CLTI patients.

ELIGIBILITY:
Inclusion Criteria:

All patients present with CLTI due to isolated infra-popliteal disease with the following criteria:

* Denovo or Recoil
* Reference tibial vessel diameter at least (2mm)
* The diseased tibial artery has a patent distal segment supplying the foot

Exclusion Criteria:

* Patients present with:

  * Previous ipsilateral infrapopliteal bypass surgery
  * Concomitant iliac or femoral artery lesion
  * Isolated pedal arch disease
  * previous atherectomy
  * Faliure to cross the lesion
  * Known hypercoagulable disorder or non-atherosclerotic vasculopathy
  * Severe renal insufficiency (eGFR <30) not on dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
• Compare the 12-month primary patency rate between the two groups. | 12 months

IPD SHARING:
Plan to Share IPD: Undecided